CLINICAL TRIAL: NCT01392274
Title: pCLE For the Diagnosis Of Cancer in Unknown Bile Duct Stricture
Acronym: FOCUS
Status: Completed | Type: Observational
Sponsor: Mauna Kea Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: MKT-2011-FOCUS
Record Dates: First submitted 2011-07-07; First posted 2011-07-12 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Cholangiocarcinoma; Bile Duct Inflammation
MeSH Terms: conditions — Cholangiocarcinoma; Cholangitis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pCLE: This trial will study only one group which will receive a standard ERCP procedure followed by pCLE

SUMMARY:
This study will collect data from patients undergoing an ERCP procedure with probe-based Confocal Laser Endomicroscopy for suspicion of bile duct cancer. the objective is to evaluate the diagnostic performance of pCLE for the diagnosis of indeterminate biliary stricture when associated with other diagnostic information (standard ERCP and tissue sampling).

DETAILED DESCRIPTION:
This trial aims at evaluating the performance diagnosis of pCLE for the detection of bile duct cancer, in patients with indeterminate biliary stricture when associated with other diagnostic information.

The hypothesis is that ERCP with Cellvizio probe-based endomicroscopy improves differentiation of biliary and pancreatic duct lesions versus ERCP alone or ERCP with tissue sampling, by improving the sensitivity of detection and by providing a real-time diagnosis.

Direct measures of accuracy (sensitivity, specificity, etc.) in the differentiation of malignant versus benign biliary duct lesions will be compared for the combination of ERCP alone, endomicroscopy plus ERCP imaging, and ERCP plus endomicroscopy plus tissue sampling. These information will be reviewed retrospectively by a second physician.

These presumptive diagnoses will be compared against a 12-month follow-up confirmed histopathologic endpoint (an initially-benign pathologic diagnosis will be confirmed by a 12-month follow-up). Secondary objectives include collecting patient management recommendation. Yet, effective management recommendation is left as the discretion of the physician.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 years of age
* Indicated for ERCP for indeterminate bile duct stricture
* Referral patients with indeterminate biliary stricture coming in for first ERCP procedure at referral institution or
* Patients who had previous non-diagnostic tissue sampling (brushing biopsies or EUS-FNA) taken during a previous ERCP or EUS-FNA for an indeterminate biliary stricture
* Willing and able to comply with study procedures and provide written informed consent to participate in the study

Exclusion Criteria:

* Subjects for whom ERCP procedures are contraindicated
* Known allergy to fluorescein dye
* Patients suffering Primary Sclerosing Cholangitis or chronic pancreatitis.
* Patients with post-transplant stricture
* If female, pregnant based on a positive hCG serum or an in vitro diagnostic test result or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Undergoing Cellvizio Endomicroscopy and Endoscopic Retrograde Cholangiopancreatography(ERCP) Imaging Procedures for Diagnosing Bile Duct Cancers
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Comparative histopathology-confirmed measures of Cellvizio endomicroscopy and ERCP accuracy in the differential diagnosis of suspicious l | 12 months
  Evaluation of pCLE diagnostic performance for the diagnosis of indeterminate biliary stricture (ie. number of patients accurately diagnosed) when associated with other diagnostic information The following calculations will be conducted: sensitivity, specificity, positive and negative predictive values, Accuracy

SECONDARY OUTCOMES:
Comparative histopathology-confirmed measures of Cellvizio endomicroscopy and ERCP accuracy in the differential diagnosis of suspicious l | 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Adam Slivka, MD, Principal Investigator — University of Pittsburh Medical Center
Locations (6):
- United States (4):
  - Yale new Haven Hospital, New Haven, Connecticut
  - New York presbyterian Weill Cornell Medical center, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington
- Institut Paoli Calmettes, Marseille, France
- Policlinico Univertitario Agostino Gemelli, Roma, Italy

REFERENCES:
- [Derived] Slivka A, Gan I, Jamidar P, Costamagna G, Cesaro P, Giovannini M, Caillol F, Kahaleh M. Validation of the diagnostic accuracy of probe-based confocal laser endomicroscopy for the characterization of indeterminate biliary strictures: results of a prospective multicenter international study. Gastrointest Endosc. 2015 Feb;81(2):282-90. doi: 10.1016/j.gie.2014.10.009. PMID 25616752